CLINICAL TRIAL: NCT00260013
Title: Transition Into Primary-care Psychiatry (TIPP): A Mental Health Demonstration Project.
Brief Title: Transition Into Primary-care Psychiatry (TIPP)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); St. Joseph's Health Care London (Other); St. Joseph's Care Group (Other)
Responsible Party: Dr. David S. Haslam, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-04-093; G03-05687 (Other Grant/Funding Number: Government of Ontario G03-05687); 10349E (Other: University of Western Ontario Research Ethics Board)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Mental Disorders
Keywords: chronic mental illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: program of care delivery

SUMMARY:
The objective of the Transition into Primary-care Psychiatry (TIPP) project is to determine how feasible it is to conduct a study to evaluate a new primary-care focused program of mental health care delivery for people with chronic mental illness. This will be done by comparing a primary-care based collaborative, interdisciplinary model to care-as-usual on health related quality of life, client symptomatology, client's perceived need of care, participant satisfaction and cost-effectiveness.

DETAILED DESCRIPTION:
The TIPP service will consist, at both the London and Thunder bay sites, of: (i) a mental health care nurse (B.Sc.N.) with at least several years experience as an outpatient mental health service clinician, and (ii) a psychiatrist with a license to practice medicine in the Province of Ontario and sensitivity to the issues of family physicians providing mental health services in the community

The TIPP intervention will involve a service delivery that is a modification of the Consultation Liaison in Primary-care Psychiatry (CLIPP) program

Four elements will act in synthesis and enable collaboration between the primary care and TIPP teams:

(i) Co-location of mental health services staff will involve the psychiatric nurse and psychiatrist visiting the family physicians' office at 1 and 3-month intervals, respectively. During these visits they will review and document the client's progress. This empowers the family physician as clinical manager. Treatment plans will be developed for family physicians that can be easily implemented. The family physician will monitor the client's status between the psychiatric nurse and psychiatrist's visits. At times of greater need, and/or impending crisis, increase in contact to every 14 days, with weekly or more from the family physician, and contacts with all providers adjusted to accommodate client needs. By developing linkages with area mental health services the psychiatric nurse will assist the family physician in co-coordinating access, while minimizing redundant use, to these services.

(ii) The TIPP nurse will select, prepare, and facilitate appropriate clients from the outpatient department for transfer to the family physician. The initial transfer process includes a face-to-face meeting with the client, TIPP nurse and family physician in family physician's office. Warning signs and symptoms of an impending relapse will allow for an opportunity for intervention to prevent or lessen the severity of a relapse. For each client a "relapse signature" strategy will be developed by the TIPP nurse to assist the family physician in detecting clients at high risk of mental illness relapse. Having obtained the client's permission significant caregivers will be routinely involved in the development and implementation of a clinical management plan. Standardized CLIPP based contact sheets\data sheets will promote efficient and effective communication between clinical care providers.

(iii) Client monitoring will be maintained by administrative staff support procedures targeted at ensuring a high level of retention and effective client follow up. The family physician will complete a Clinical Global Impression Scale (CGIS) (severity and change scores) every 3 months in the first year then at each visit for the remainder of the project. The CGIS will not add time to the clinical time with the clients. An administrative member of the project receiving these scales will alert the appropriate clinical providers for clients whose condition is not improving as judged by the family physician.

(iv) Telephone back up for the family physicians' whose clients are involved in the project will be provided by a project psychiatrist and/or psychiatric nurse.

The outcomes of the TIPP intervention clients will be compared to those who receive post outpatient service transfer care-as-usual from their family physician. The clients in this group will obtain any and all services normally available inside or outside their primary care service, including re-referral to specialty mental health care. No additional services will be provided for the care-as-usual group, but no usual services will be limited or withheld. Design features to ensure the interests of the control group are considered include outcomes assessment for both groups at 6, and 12 months, as well as at the projects end point. Should significant clinical concerns be noted by the rater during the assessment a systematic process will allow for the family physician to be notified so as to minimize the risk of compromised care.

ELIGIBILITY:
Inclusion Criteria:

* (1) receiving outpatient psychiatric clinic services through the St. Joseph's Care Group Lakehead Psychiatric Hospital in the Community Mental Health Services program, Thunder Bay, Ontario or at the Regional Mental Health Care, Specialized Adult Service, London, Ontario 2) 18-65 years of age; 3) chronic moderate to severe mental illness - all scores below severe or very severe rating on the Threshold Assessment Grid; 4) duration of mental illness of at least 2 years; 5) not regularly receiving psychiatric or mental health care from another family physician, and; 6)capable of understanding the nature of the project and can give consent.

Exclusion Criteria:

* Clients will be excluded if at the time of recruitment they:

  1. have an unstable mental illness;
  2. had a psychiatric hospitalization admission within the last past 6 months;
  3. used crisis intervention within the past 6 months (requiring subsequent contact greater than once per week);
  4. had a history of self-harm over the past 6 months;
  5. had a history of harm to others over the past 6 months;
  6. had drug and alcohol problems over the past 6 months that would contribute significantly to clinical destabilization;
  7. have unmet major psychosocial needs (including homelessness and marked poverty), and;
  8. are experiencing a serious medical illness that is unstable and that contributes to instability of mental illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Quality of Well Being

SECONDARY OUTCOMES:
Symptomatology
Perceived need for care
Satisfaction
Cost Effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: David RS Haslam, MSc MD FRCPC, Principal Investigator — St. Joseph's Health Care London; John M Haggarty, BSc MD FRCPC, Principal Investigator — St. Joseph's Care Group
Locations (1):
- St. Joseph's Care Group Lakehead Psychiatric Hospital, Thunder Bay, Ontario, Canada